CLINICAL TRIAL: NCT00830843
Title: Inhalatorial Sedation in Patient With SAH Versus Conventional Intravenous Sedation (GAS-SAH)
Brief Title: Inhalatorial Sedation in Patient With Subarachnoid Hemorrhage (SAH) Versus Conventional Intravenous Sedation
Acronym: GAS-SAH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Prof. Giuseppe Citerio, MD, Azienda Ospedaliera San Gerardo di Monza
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1-citerio
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2011-11

CONDITIONS: Stroke; Subarachnoid Hemorrhage
Keywords: SAH; sedation; anesthesia
MeSH Terms: conditions — Stroke; Subarachnoid Hemorrhage | interventions — Propofol; Isoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): Propofol(3-4 mg/kg/ora)administrated for 2 hours.
  Interventions: Drug: Propofol
- Isoflurane (Experimental): Isoflurane inhalatorial administration for 2 hours at 0.8-1.0% Minimum Alveolar Concentration
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Propofol — Propofol(3-4 mg/kg/ora)administrated for 2 hours.
  Other Names: Diprivan
  Arms: Propofol
Drug: Isoflurane — Isoflurane inhalatorial administration for 2 hours at 0.8-1.0% Minimum Alveolar Concentration
  Arms: Isoflurane

SUMMARY:
Recent study has shown that inhalatory sedation is a practicable, effective and not risky method in Intensive Care Unit. Sevoflurane effect on cerebral system have been described in previous studies: it causes an increasing of cerebral blood flow and a decrease of oxygen cerebral consumption. Clinical strategy for Subarachnoid Hemorrhage is orientated to increase cerebral blood flow to limit vasospasm phenomena after SAH. Scope of this study is to evaluate the Cerebral Blood Flow variation associated to Isoflurane sedation versus conventional sedation with propofol .

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of aSAH
* indication to DVE positioning
* clinical indication to sedation and assisted ventilation
* indication to ICP and CBF monitoring
* age > 18

Exclusion Criteria:

* documented cranial hypertension (ICP>18) not controller by liquor drainage
* age < 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow | after 2 hours of drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Federico Villa, MD, Principal Investigator — Azienda Ospedaliera San Gerardo Monza
Locations (1):
- Azienda Ospedaliera San Gerardo, Monza, Monza, Italy

REFERENCES:
- [Background] Newberg LA, Milde JH, Michenfelder JD. The cerebral metabolic effects of isoflurane at and above concentrations that suppress cortical electrical activity. Anesthesiology. 1983 Jul;59(1):23-8. doi: 10.1097/00000542-198307000-00005. PMID 6859608
- [Background] Maekawa T, Tommasino C, Shapiro HM, Keifer-Goodman J, Kohlenberger RW. Local cerebral blood flow and glucose utilization during isoflurane anesthesia in the rat. Anesthesiology. 1986 Aug;65(2):144-51. doi: 10.1097/00000542-198608000-00003. PMID 3740503
- [Background] Reinstrup P, Ryding E, Algotsson L, Messeter K, Asgeirsson B, Uski T. Distribution of cerebral blood flow during anesthesia with isoflurane or halothane in humans. Anesthesiology. 1995 Feb;82(2):359-66. doi: 10.1097/00000542-199502000-00006. PMID 7856894
- [Background] Zhao P, Peng L, Li L, Xu X, Zuo Z. Isoflurane preconditioning improves long-term neurologic outcome after hypoxic-ischemic brain injury in neonatal rats. Anesthesiology. 2007 Dec;107(6):963-70. doi: 10.1097/01.anes.0000291447.21046.4d. PMID 18043065
- [Background] Zhao P, Zuo Z. Isoflurane preconditioning induces neuroprotection that is inducible nitric oxide synthase-dependent in neonatal rats. Anesthesiology. 2004 Sep;101(3):695-703. doi: 10.1097/00000542-200409000-00018. PMID 15329594
- [Background] McAuliffe JJ, Joseph B, Vorhees CV. Isoflurane-delayed preconditioning reduces immediate mortality and improves striatal function in adult mice after neonatal hypoxia-ischemia. Anesth Analg. 2007 May;104(5):1066-77, tables of contents. doi: 10.1213/01.ane.0000260321.62377.74. PMID 17456654
- [Background] Zheng S, Zuo Z. Isoflurane preconditioning induces neuroprotection against ischemia via activation of P38 mitogen-activated protein kinases. Mol Pharmacol. 2004 May;65(5):1172-80. doi: 10.1124/mol.65.5.1172. PMID 15102945
- [Background] Lee JJ, Li L, Jung HH, Zuo Z. Postconditioning with isoflurane reduced ischemia-induced brain injury in rats. Anesthesiology. 2008 Jun;108(6):1055-62. doi: 10.1097/ALN.0b013e3181730257. PMID 18497606
- [Background] Kapinya KJ, Lowl D, Futterer C, Maurer M, Waschke KF, Isaev NK, Dirnagl U. Tolerance against ischemic neuronal injury can be induced by volatile anesthetics and is inducible NO synthase dependent. Stroke. 2002 Jul;33(7):1889-98. doi: 10.1161/01.str.0000020092.41820.58. PMID 12105371
- [Background] L'her E, Dy L, Pili R, Prat G, Tonnelier JM, Lefevre M, Renault A, Boles JM. Feasibility and potential cost/benefit of routine isoflurane sedation using an anesthetic-conserving device: a prospective observational study. Respir Care. 2008 Oct;53(10):1295-303. PMID 18811990
- [Background] Berton J, Sargentini C, Nguyen JL, Belii A, Beydon L. AnaConDa reflection filter: bench and patient evaluation of safety and volatile anesthetic conservation. Anesth Analg. 2007 Jan;104(1):130-4. doi: 10.1213/01.ane.0000248221.44383.43. PMID 17179257
- [Background] Sackey PV, Martling CR, Nise G, Radell PJ. Ambient isoflurane pollution and isoflurane consumption during intensive care unit sedation with the Anesthetic Conserving Device. Crit Care Med. 2005 Mar;33(3):585-90. doi: 10.1097/01.ccm.0000156294.92415.e2. PMID 15753751
- [Background] Sackey PV, Martling CR, Granath F, Radell PJ. Prolonged isoflurane sedation of intensive care unit patients with the Anesthetic Conserving Device. Crit Care Med. 2004 Nov;32(11):2241-6. doi: 10.1097/01.ccm.0000145951.76082.77. PMID 15640636
- [Derived] Villa F, Iacca C, Molinari AF, Giussani C, Aletti G, Pesenti A, Citerio G. Inhalation versus endovenous sedation in subarachnoid hemorrhage patients: effects on regional cerebral blood flow. Crit Care Med. 2012 Oct;40(10):2797-804. doi: 10.1097/CCM.0b013e31825b8bc6. PMID 22824929